CLINICAL TRIAL: NCT00352651
Title: Placebo-Controlled Study of Pregabalin for the Pain of Acute Herpes Zoster
Brief Title: Study to Find Out if Therapy With the Drug Pregabalin Relieves Pain During Shingles Compared With Placebo
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This study should be terminated as the study has been closed for years and the investigator has since retired. No records are available.
  Thank you, Marlene
Sponsor: University of California, San Francisco (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Michael Rowbotham, University of California, San Francisco
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: H11609-27650
Record Dates: First submitted 2006-07-12; First posted 2006-07-14 (Estimated); Last update posted 2011-04-14 (Estimated); Status verified 2011-03

CONDITIONS: Herpes Zoster; Postherpetic Neuralgia
Keywords: Acute Herpes Zoster (AHZ); Postherpetic Neuralgia (PHN); Pregabalin; Lyrica; Pain
MeSH Terms: conditions — Herpes Zoster; Neuralgia, Postherpetic; Pain | interventions — Pregabalin

INTERVENTIONS:
Drug: Pregabalin

SUMMARY:
The purpose of this study is to see if therapy with the drug pregabalin relieves pain during shingles compared with placebo. A placebo is an inactive substance. Pregabalin is a drug marketed as Lyrica™ in the United States for the treatment of seizures, diabetic neuropathy, and post-herpetic neuralgia. The use of pregabalin and drugs like it for the treatment of pain during the acute phase of shingles is experimental. Thirty four subjects will complete the study at the University of California, San Francisco (UCSF) Pain Clinical Research Center. This study is funded by Pfizer Global Research.

DETAILED DESCRIPTION:
The varicella zoster virus (VZV) is the smallest of the double-stranded DNA herpes viruses, and the only one capable of producing two different diseases, varicella (chickenpox) and herpes zoster (acute herpes zoster [AHZ], shingles). The incidence of AHZ, and the secondary VZV infection, is strongly age-dependent and reaches 1% per year by age 80 and there are between 300,000 and 1 million new cases of AHZ each year in the US. AHZ is almost always painful, and the pain can be of disabling severity, rendering some sufferers bed-bound and too incapacitated to carry out normal activities, leading to weight loss and dehydration sufficient to require inpatient therapy. The elderly are especially likely to suffer severe pain.

The most common complication of AHZ is development of postherpetic neuralgia (PHN). Although the overall incidence of PHN after AHZ is about 10%, the incidence has been reported to rise as high as 80% in those over the age of 80. In all published studies, age and greater severity of initial zoster pain are each found to significantly increase the risk of developing PHN. Severe zoster pain is believed to correlate with a more severe cutaneous outbreak, more severe inflammation of the nerve trunk, and possibly greater injury to primary afferent nerve fibers.

There are two separate issues to address when discussing the pain of AHZ. The first is managing the AHZ pain itself, because the burden of suffering is so high. The second is reducing the incidence of PHN. Both issues need to be considered in trial design, in part because severe AHZ pain is itself a risk factor for PHN. Studies of the analgesic effect of pregabalin suggest an analgesic profile similar to that of gabapentin. We would therefore predict, that pregabalin would reduce the pain associated with AHZ and possibly prevent development of PHN.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 21 years of age or older
2. Subjects must have an acute outbreak of herpes zoster (HZ) with unilateral skin rash and pain; the diagnosis will be based on physical examination and review of available medical records confirming the outbreak.
3. Subjects must have had pain present for more than 3 days but less than 42 days after onset of the herpes zoster skin rash.
4. Subjects at screening must have an average score of at least 40 mm on the visual analog scale (VAS) of the SF-McGill Pain Questionnaire.
5. Subjects must weigh more than 110 pounds and have a body mass index greater than or equal to 20.
6. No medications for AHZ pain other than nonsteroidal anti-inflammatory drugs (NSAIDs), acetaminophen and opioids; maintained at a stable dose throughout the study.
7. No use of topical medications less than 12 hours prior to each study medication visit. No use of NSAIDs, acetaminophen, or opioids less than 2 hours prior to each study medication visit.
8. Ability to understand and follow the instructions of the investigator, including completion of the study diaries as described in the protocol.
9. Ability to provide informed written consent.

Exclusion Criteria:

1. The AHZ outbreak is complicated by stroke or myelopathy.
2. Patients with signs of spinal cord or brainstem injury from HZ.
3. Subjects who have demonstrated a hypersensitivity to pregabalin (or gabapentin) or who have been previously treated with either.
4. Subjects who have undergone neurolytic or neurosurgical therapy for AHZ.
5. Subjects treated with local anesthetic nerve blocks within 48 hours of study entry.
6. Subjects with a creatinine clearance of 60 mL/minute or less or significant renal disease as determined by study physician.
7. Clinically significant hepatic, respiratory, hematological, cardiovascular or neurological disease.
8. Subjects having other severe pain that may confound assessment of the AHZ pain.
9. Subjects who have serious, unstable, or clinically significant medical or psychological conditions, which, in the opinion of the investigator(s), would compromise the subject's participation in the study (including clinically significant dehydration or unstable vital signs).
10. Subjects taking or having taken any other experimental drugs, drugs not approved in the United States, or participating in or having participated in other clinical studies in the 30 days prior to this clinical trial.
11. Pregnant or lactating women.
12. Subjects who are currently taking anticonvulsants.
13. Subjects who have a history of illicit drug or alcohol abuse within the last year.
14. Subjects who are considered unreliable as to medication compliance or adherence to scheduled appointments, or for other reasons are felt to be inappropriate for inclusion in the study as determined by the investigators.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2006-06; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Subjects' pain ratings using the visual analog scale (VAS) (0-100 mm) from pre-drug through 6 hours post-drug

SECONDARY OUTCOMES:
Subject ratings of allodynia severity to 3 strokes with a foam brush, the surface areas of greatest pain and allodynia, side effect scores, and a Category Pain Relief Scale rating from 0 (pain worsened) to 5 (complete pain relief)

CONTACTS AND LOCATIONS:
Overall Officials: Karin L. Petersen, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Pain Clinical Research Center, San Francisco, California, United States

REFERENCES:
- [Derived] Jensen-Dahm C, Rowbotham MC, Reda H, Petersen KL. Effect of a single dose of pregabalin on herpes zoster pain. Trials. 2011 Feb 28;12:55. doi: 10.1186/1745-6215-12-55. PMID 21356040